CLINICAL TRIAL: NCT00149630
Title: Effectiveness of Disulfiram for Treating Cocaine Dependence in Individuals With Different Dopamine Beta Hydroxylase (DBH) Genes
Brief Title: Pharmacogenetics of Disulfiram for Cocaine
Acronym: Disulfiram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Yale University (Other)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-18197-2; P50DA018197-02 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Cocaine Dependence; Opioid Dependence
Keywords: Opioid Dependence; Substance Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders | interventions — Disulfiram; Methadone; Cognitive Behavioral Therapy; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disulfiram, Methadone (w/lactose) & CBT (Experimental): Participants are randomly assigned to receive a daily dose of 250 mg of disulfiram for 12 weeks, while concurrently receiving methadone treatment. All participants will stop receiving study medication at week 14, at which point they will undergo a 4-week methadone detoxification period.
  Interventions: Drug: Disulfiram; Drug: Methadone; Behavioral: CBT; Other: Lactose
- Placebo, Methadone (w/lactose) & CBT (Active Comparator): Participants are randomly assigned to receive a daily dose of a sugar pill to mimic the experimental drug disulfiram for 12 weeks, while concurrently receiving methadone treatment. All participants will stop receiving all medication at week 14, at which point they will undergo a 4-week methadone detoxification period.
  Interventions: Drug: Methadone; Behavioral: CBT; Other: Lactose

INTERVENTIONS:
Drug: Disulfiram — Disulfiram 250 mg/day by mouth daily during study weeks 2-13. Disulfiram discontinued during study weeks 14-15.
  Other Names: Antabuse
  Arms: Disulfiram, Methadone (w/lactose) & CBT
Drug: Methadone — Initial dose 25 mg; increased by 5 mg at each subsequent daily dosing until 60 mg maintenace dose reached.
  Other Names: Symoron; Dolophine; Amidone; Methadose; Physeptone; Heptadon
Behavioral: CBT — 1-hour weekly, individual, manual-guided Cognitive Behaviorial Therapy.
  Other Names: Cognitive Behavioral Therapy
Other: Lactose — Lactose was added to both the active disulfiram and placebo doses so they tasted identical.
  Other Names: lactose suspension

SUMMARY:
Previous research has shown that disulfiram, a medication sometimes used for treating alcoholism, discourages cocaine use among cocaine addicts who are undergoing methadone treatment. By blocking the enzyme dopamine beta hydroxylase (DBH), disulfiram increases levels of dopamine and produces an unpleasant sense of hyperstimulation and discomfort in cocaine users. This study will evaluate the effectiveness of disulfiram in preventing drug relapse among cocaine and opiate addicts with varying inherited levels of DBH.

DETAILED DESCRIPTION:
Dopamine, a type of neurotransmitter, is the brain's "feel good" chemical. The amount of dopamine in the body may be an important factor in how cocaine addicts respond to treatment. Disulfiram, like cocaine, enhances dopamine activity. Upon taking disulfiram, subsequent intake of cocaine may elevate dopamine to excessive levels that produce extreme discomfort. DBH is an enzyme that breaks down dopamine. A particular variation in the DBH gene can affect the amount of dopamine that is released in the body. Therefore, cocaine addicts with varying DBH genes may respond differently to treatment. The purpose of this study is to compare the effectiveness of disulfiram in preventing relapse among methadone-maintained individuals addicted to both cocaine and opioids who may have different DBH genes.

This 17-week study will begin with a 2-week methadone stabilization period. Participants will then be randomly assigned to receive a daily dose of either 250 mg of disulfiram or placebo for 12 weeks, while concurrently receiving methadone treatment. All participants will stop receiving study medication at Week 14, at which point they will undergo a 4-week methadone detoxification period. Participants will report cocaine and other drug use, as well as any cocaine cravings that they experience. Cocaine levels will be monitored throughout the study with urine tests. The DBH gene of each participant will be examined to determine its specific make-up and any particular variations.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for opioid dependence, as determined by documentation of prior treatment for addiction; signs of withdrawal; self-reported history of dependence for at least 1 year; and a positive urine test for opioids
* Meets DSM-IV diagnosis criteria for cocaine dependence, as determined by self-reported use of cocaine at least once weekly for at least 1 month prior to study entry; a positive urine test for cocaine; and a score greater than 3 on the Severity Dependence Scale
* If female, willing to use contraception throughout the study

Exclusion criteria:

* Meets DSM-IV diagnosis criteria for dependence on any drugs other than opiates, cocaine, or tobacco
* Current major psychiatric illness, including schizophrenia, bipolar disorder, or other psychotic disorder
* Current suicidal or homicidal ideation
* Current use of a prescribed psychotropic medication that cannot be discontinued
* History of or current major medical illness, including major heart, kidney, endocrine, or liver disorder; abnormal liver function (SGOT or SGPT levels three times greater than normal);
* High risk factor for heart disease, seizure disorders, or any illness for which disulfiram or methadone treatment would be inadvisable
* Currently taking metronidazole or clotrimazole
* Pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas PS Jr, Nielsen EM, Spellicy CJ, Harding MJ, Ye A, Patriquin M, Hamon SC, Kosten TR, Nielsen DA. The OPRD1 rs678849 variant influences outcome of disulfiram treatment for cocaine dependency in methadone-maintained patients. Psychiatr Genet. 2021 Jun 1;31(3):88-94. doi: 10.1097/YPG.0000000000000279. PMID 33953123
- [Derived] Spellicy CJ, Kosten TR, Hamon SC, Harding MJ, Nielsen DA. The MTHFR C677T Variant is Associated with Responsiveness to Disulfiram Treatment for Cocaine Dependency. Front Psychiatry. 2013 Jan 14;3:109. doi: 10.3389/fpsyt.2012.00109. eCollection 2012. PMID 23335901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 74 opioid and cocaine dependent subjects were drawn from a sample of 93 candidates who entered into a 2-week screening period for stabilization on methadone maintenance between 2005 and 2006 at Yale University (n=40) and then from between 2006 and 2008 at Baylor College of Medicine (n=53).
Pre-assignment Details: Eleven subjects were excluded prior to randomization because they did not have at least one urine toxicology positive for opiates or cocaine metabolites during the two-week screening. Another eight subjects were lost to follow-up prior to randomization.
Groups:
- Disulfiram: 250 mg/day with methadone daily during study weeks 2-13. Medication will be discontinued during study weeks 14-15.
- Placebo: Inactive medication (placebo) with methadone daily during study weeks 2-13. Inactive medication will be discontinued during study weeks 14-15.
Period: Overall Study
Arm/Group | Disulfiram | Placebo
Started | 34 | 40
Completed | 26 | 35
Not Completed | 8 | 5
Not completed — Incarceration | 2 | 0
Not completed — Treatment Programs | 4 | 5
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disulfiram | Placebo | Total
Number analyzed (Participants) | 34 | 40 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 40 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.5) | 40 (10) | 38.75 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 24 | 28 | 52
Region of Enrollment [Number; unit: participants]
  United States | 34 | 40 | 74

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology for Cocaine.
Time Frame: Thrice weekly, baseline through week 14.
Population: 74 cocaine and opioid-codependent (DSM-V) subjects were stabilized on methadone for 2 weeks and subsequently randomized into disulfiram (250mg/day, n=34) and placebo groups (n=40) for 10 weeks. We genotyped the DBH gene polymorphism that reduces DBH enzyme levels and evaluated its role for increasing cocaine free urines with disulfiram.
Measure: Mean (Standard Error); unit: % cocaine + urines over 2 week blocks
Groups:
- Placebo CC: Subjects who received placebo with a genotype of CC.
- Placebo CT/TT: Subjects who received placebo with genotype CT/TT.
- Disulfiram CC: Subjects who received Disulfiram with genotype CC.
- Disulfiram CT/TT: Subjects who received Disulfiram with genotype CT/TT.
Arm/Group | Placebo CC | Placebo CT/TT | Disulfiram CC | Disulfiram CT/TT
Number analyzed (Participants) | 21 | 19 | 17 | 17
% cocaine + urines over 2 week blocks | 84 (5) | 68 (5) | 56 (5) | 67 (5)

2. Secondary Outcome: Retention by Treatment Condition.
Description: Treatment retention for full 12 weeks of study.
Time Frame: 12 weeks
Population: 74 cocaine and opioid-codependent(DSM-V)subjects were stabilized on methadone for 2 weeks and subsequently randomized into disulfiram (250 mg/day, n=34) and placebo groups (n=40) for 10 weeks. We genotyped the DBH gene polymorphism that reduced DBH enzyme levels and evaluated its role for increasing cocaine free urines with disulfiram.
Measure: Number; unit: % of subjects who complete 12 wks study
Arm/Group | Disulfiram | Placebo
Number analyzed (Participants) | 34 | 40
% of subjects who complete 12 wks study | 77 | 87

ADVERSE EVENTS:
Groups:
- Disulfarim: 250 mg/day with methadone daily during study weeks 2-13. Study medicine discontinued during study weeks 14-15.
- Placebo: Inactive medicine (placebo)with methadone during study weeks 2-13. Inactive medicine discontinued during study weeks 14-15.
Arm/Group | Disulfarim | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/40
Other Adverse Events (participants affected / at risk) | 3/34 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disulfarim (N=34) | Placebo (N=40)
Reduced sexual functioning. (Renal and urinary disorders) | 1 (1) | 0 (0) — One disulfiram patient left the study for reduced sexual functioning but this was considered as related to the methadone.
Suicide gesture. (Psychiatric disorders) | 0 (0) | 1 (1) — One placebo patient made suicidal gesture of superficially cutting his wrist but was not hospitalized and completed 12 weeks.
Arm numbness. (Vascular disorders) | 1 (1) | 0 (0) — Disulfiram patient had arm numbness that resolved spontaneously during the trial without any changes in medication. Patient completed 12 weeks of trial.
Arm numbness and back rash. (Vascular disorders) | 1 (1) | 0 (0) — Disulfiram patient had arm numbness and back rash and left at Week 6.

LIMITATIONS AND CAVEATS:
The sample size is small for this genetic association study, and larger replications of this preliminary study are needed. Most cocaine abusers are not also opioid dependent, which limits generalization of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes